CLINICAL TRIAL: NCT06033625
Title: Joint Awareness After Cemented or Cementless Total Knee Replacement: Does it Change?
Brief Title: Joint Awareness After Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, İsmail Demirkale, Clinical professor, Saglik Bilimleri Universitesi
Other Study IDs: 2470
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis; Arthroplasty Complications
Keywords: Joint Awareness; Total Knee Replacement; Cementless; Forgotten Joint Score; Patient's Joint Perception
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cd-TKR: Bicompartmental cemented cruciate retaining Total knee replacement
- Cs-TKR: Bicompartmental cementless cruciate retaining Total knee replacement
  Interventions: Procedure: CEMENTLESS TOTAL KNEE REPLACEMENT

INTERVENTIONS:
Procedure: CEMENTLESS TOTAL KNEE REPLACEMENT — CEMENTLESS CRUCIATE RETAINING BICOMPARTMENTAL TOTAL KNEE REPLACEMENT
  Groups: Cs-TKR

SUMMARY:
Total knee replacement (TKR) is accepted as treatment of choice for end stage gonarthrosis. It is performed cemented or cementless and although cemented implants were shown to decrease bone density more than cementless fixations there is no evidence-based difference between them in the literature. As far as the investigators are concerned, the effect of cementation on patients' joint perception has never been studied so far.

DETAILED DESCRIPTION:
In this longitudinal case-control study, joint awareness in prosthetic reconstruction was evaluated in 150 knees (75 cemented TKR, 75 cementless TKR) of 136 patients. They were operated between 2015 and 2017 in our institution with minimum 5 years of follow up. All the patients in each group were operated by two senior surgeons that were experienced for more than 10 years in arthroplasty. To reduce selection bias, logistic regression was used to develop propensity-matched pairs based on gender, age, body mass index (BMI), preoperative coronal plane deformity, preoperative range of motion (ROM) and appropriateness for TKA indication. Demographic and clinical data including sex, age and time since surgery were collected. The subjects' joint perception and the WOMAC clinical scores were recorded and compared. Joint awareness is assessed with Forgotten Joint Score (FJS) which has 12 questions and with Patient's Joint Perception questionnaire (PJP) which is a single question with 5 possible answers, rating from the highest expected result "like a native or natural joint" to the worse possible case "a non-functional joint". Other than clinical scores, laboratory parameters, blood transfusion needs, tourniquet time, complications (septic/aseptic loosening, periprosthetic fracture, instability) and revision rates were also compared.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* "appropriate'' TKA indication according to Modified Escobar System

Exclusion Criteria:

* secondary osteoarthritis
* previous surgery to the knee
* valgus knee
* uncontrolled diabetes

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with primary end stage varus osteoarthritis of the knee
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Forgotten Joint Score-12 (FJS-12) | 1 year after index surgery and at the end of 5th year
  a patient-reported outcome measure intended to determine a patient's ability to "forget" about their affected joint after surgery or treatment and uses a 5-point Likert response format (0, never; 1, almost; 2, seldom; 3,sometimes; and 4, mostly) with high scores indicate good outcome, which means a high degree of "forgetting" the joint
Patient's Joint Perception questionnaire (PJP) | 1 year after index surgery and at the end of 5th year
  The PJP is a single question with 5 possible answers, rating from the highest expected result "like a native or natural joint" to the worsening gradually as Artificial joint with no restriction, Artificial joint with minimal restriction, Artificial joint with major restriction and "a non-functional joint"

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 1 year after index surgery and at the end of 5th year
  The WOMAC is a specific, valid, and reliable measure for OA, consisting of 24 questions in three subcategories: pain, stiffness, and physical function. Each question is scored using a Likert scale as follows: 0=nothing, 1=mild, 2=moderate, 3=severe, 4=very severe. The score for each section is calculated separately, and the total score ranges from 0 to 100. Higher scores indicate an increase in pain and stiffness, as well as a deterioration in physical function.